CLINICAL TRIAL: NCT05328830
Title: Comparison of the Effects of Instrumental Assisted Soft Tissue Mobilization and Foam Roller on Delayed Muscle Pain.
Brief Title: Soft Tissue Mobilization Effects on Doms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Erdoğan Çetintaş, principal investigator, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ETK00-2021-0070
Record Dates: First submitted 2022-01-05; First posted 2022-04-14 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Performance
Keywords: doms; muscle strength; flexibility; recovery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Instrument assisted soft tissue mobilization group (Experimental): Instrument assisted soft tissue mobilization will be applied after 30 minutes of DOMS creation
  Interventions: Other: Instrument assisted soft tissue mobilization
- Foam roller (Experimental): Foam roller will be applied after 30 minutes of DOMS creation
  Interventions: Other: Foam Roller
- control group (No Intervention): no intervention

INTERVENTIONS:
Other: Instrument assisted soft tissue mobilization — Myofascial release technique will be applied to the Quadriceps, Hamstring and Gastrocnemius muscles of the participant's dominant lower extremity with the Graston technique®. The application will be at 450 angles for each muscle, 2 minutes, for a total of 6 minutes. The IASTM application will include sweep-fan-sweep strokes and cycle through each muscle for the specified time.
  Arms: Instrument assisted soft tissue mobilization group
Other: Foam Roller — Will be applied to the Quadriceps, Hamstring and Gastrocnemius muscles of the participant's dominant lower extremity using rigid Foam Roller. A total of 6 minutes will be applied to a person, 2 minutes for each muscle. Pressure intensity; According to the Visual Analog Scale, which is the point where pain will not be felt but moderate to severe discomfort will be felt, it will be done at a severity of 7/10.
  Arms: Foam roller

SUMMARY:
Aim: The aim of the study was to examine and compare the time-dependent effects of IASTM and FR applications on delayed muscle pain and physical performance.

Method: 50 physically active healthy male individuals between the ages of 20-35 will be included in the study. Participants will be divided into 3 separate groups as instrument assisted soft tissue mobilization(IASTM), foam roller (FR) and control group. DOMS creation protocol will be implemented after preliminary evaluation. IASTM and FR groups will be treated after the formation of doms. The control group will not be applied. participants are evaluated 1 day before the doms were created and at 24, 48 and 72 hours after doms created. Subjetcs were tested for physical activity level with IPAQ-SF, flexibility with sit and reach test, pain with Visual analog scale, edema with thigh circumference measurement, explosive power with horizontal and vertical jump test, dynamic balance with y balance test and isokinetic muscle strength of the quadriceps and hamstring muscles with isokinetic dynamometer.

DETAILED DESCRIPTION:
Muscle soreness after exercise is often referred to as delayed onset muscle soreness (DOMS). DOMS is common in people who do strenuous and unusual exercise and physical activity. DOMS, also called Grade 1 muscle strain, is characterized by localized tenderness and pain. DOMS typically peaks between 24-72 hours after strenuous exercise and disappears within 5-7 days.2-4 Associated with exercises involving eccentric muscle movement DOMS also affects athletic performance by causing decreased range of motion and reduced peak torque.

According to literature, many improvement strategies have been used by athletes, coaches and health professionals to minimize DOMS symptoms and improve performance. These strategies include massage, stretching exercises and the use of anti-inflammatory drugs. Studies conducted in different populations to date show that the results of these treatments on DOMS usually have minimal analgesic effects. Improvements in strength and flexibility have also been observed in some studies.

Myofascial release method, developed by James Cyriax, Instrument assisted soft tissue mobilization (IASTM) is applied with specially designed instruments. In particular, the use of instruments in the technique, which has been shown to have a mobilizing effect on soft tissue to reduce pain, increase range of motion and function, creates a deeper effect and allows specific treatment. It is also known to provide a mechanical advantage for the clinician by reducing the pressure on the hand. Current studies show that IASTM can improve joint ROM change the perception of pain and increase local circulation

Foam Roller (FR), another method used for myofascial relaxation, is a method that has been frequently researched in recent years, especially in the warming and recovery phases. FR includes a wide variety of therapy techniques, including massage and self-massage. Myofascial release is used to treat somatic dysfunction causing pain and limitation. Self myofascial release is performed using FR or stick. To demonstrate the effect of self-myofascial relaxation, studies focused on the effect of FR on increasing ROM, reducing muscle soreness, and lower extremity biomechanical performance. The first effect is associated with recovery and recovery, while the second effect is associated with performance. There are several studies reporting that FR also has a major impact on improving flexibility. In fact, there are studies reporting that it shows this effect even after a single FR session.

The number of studies investigating or comparing the effects of FR and IASTM techniques on delayed muscle pain is very limited in the literature. Studies comparing the effects of the two techniques have generally compared their effectiveness in the upper extremity muscles. In the lower extremity, there is only one study investigating and comparing the effects of both treatment methods in healthy active individuals. In this study, only the effects of techniques on flexibility were evaluated. Therefore, the aim of our study is to examine and compare the time-dependent effects of IASTM and FR applications on delayed muscle pain and physical performance.

Method:

Participants who want to take part in the study will first be informed about the study in written and verbal form and their written consent will be obtained. Then, the socio-demographic characteristics and information of all participants will be recorded. On the same day, the assessments detailed below will be audited by all participants and they will be given the opportunity to practice in order to adapt to the assessment methods. Preliminary evaluations of all participants (all evaluations mentioned in the evaluations section) will be taken at least 48 hours after the practice day. After the preliminary evaluations, individuals will be randomly divided into 3 groups with GraphPad - version 8.4.3 software in order to determine which group (foam roller/instrument assisted soft tissue mobilization or control group) the participants will be in. Treatment methods to be applied to the groups were divided into two as IASTM and Foam roller.

Group 1 (Foam Roller): It will be applied to the Quadriceps, Hamstring and Gastrocnemius muscles of the participant's dominant lower extremity using a rigid FR. A total of 6 minutes will be applied to a person, 2 minutes for each muscle. Pressure intensity; According to the Visual Analogue Scale, which is the point where pain will not be felt but moderate to severe discomfort will be felt, it will be done at a severity of 7/10.

Group 2 (IASTM): Myofascial release technique will be applied to the Quadriceps, Hamstring and Gastrocnemius muscles in the dominant lower extremity of the participant with the Graston technique®, the instrument to be used in this technique. The application will be at 45° angles for each muscle, 2 minutes, for a total of 6 minutes. The IASTM application will include sweep-fan-sweep strokes and cycles will be performed along each muscle for a specified time.

Group 3 (control): Individuals in this group will be asked not to participate in any physical activity during the evaluations (5 days) and to do their normal daily activities

Method: After the first evaluations, DOMS will be applied 48 hours later. Immediately after the DOMS is created, FR will be applied to those in Group 1, IASTM will be applied to those in Group 2, and no application will be made to those in Group 3. On the same day, 30 minutes after the applications, pain (VAS) and edema (Quadriceps circumference measurement) will be evaluated. At 24, 48 and 72 hours, all evaluations will be repeated to the participants.

DOMS creation protocol: It will be created by eccentric contraction in the isokinetic device. The patient will be positioned with the knee at 90° flexion. Then, the knee extensors will be asked to perform 5 sets of 15 repetitions of maximal voluntary eccentric contraction at an angular speed of 60°/s. There will be 2 minutes of rest between sets.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active (who do moderate-vigorous physical activity at least 2 times a week)
* Those who are moderately and/or highly active according to the IPAQ scale
* Between the ages of 20-35
* Doing moderate to severe physical activity at least 2 times a week
* Those who have not received IASTM or Foam Roller application in the last 30 days

Exclusion Criteria:

* Those who are allergic to the intermediate used material in IASTM application
* Those who use alcohol and supplements
* Those who have any lower extremity injury in the last 6 months
* Those with orthopedic or neurological disease

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 42 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
change between baseline of pain assessment and immidiately after DOMS created. | Assessments will be performed on baseline and immdidiately after DOMS created.
  Visual Analog Scale will be used for pain assessment.
change between baseline of pain assessment and 1 day after DOMS created. | Assessments will be performed on baseline and 1 day after DOMS created.
  Visual Analog Scale will be used for pain assessment.
change between baseline of pain assessment and 2 days after DOMS created. | Assessments will be performed on baseline and 2 days after DOMS created.
  Visual Analog Scale will be used for pain assessment.
change between baseline of pain assessment and 3 days after DOMS created. | Assessments will be performed on baseline and 3 days after DOMS created.
  Visual Analog Scale will be used for pain assessment.

SECONDARY OUTCOMES:
change between baseline of flexibility test and 1 day after DOMS created. | Assessments will be performed on baseline and 1 day after DOMS created.
  sit and reach test will be used for flexility assessment
change between baseline of flexibility test and 2 days after DOMS created. | Assessments will be performed on baseline and 2 days after DOMS created.
  sit and reach test will be used for flexility assessment
change between baseline of flexibility test and 3 days after DOMS created. | Assessments will be performed on baseline and 3 days after DOMS created.
  sit and reach test will be used for flexility assessment
change between baseline of muscle strength test and 1 day after DOMS created. | Assessments will be performed on baseline and 1 day after DOMS created.
  Isokinetic dynamometer will be used for muscle strength assessment
change between baseline of muscle strength test and 2 days after DOMS created. | Assessments will be performed on baseline and 2 days after DOMS created.
  Isokinetic dynamometer will be used for muscle strength assessment
change between baseline of muscle strength test and 3 days after DOMS created. | Assessments will be performed on baseline and 3 days after DOMS created.
  Isokinetic dynamometer will be used for muscle strength assessment
change between baseline of vertical jump test and 1 day after DOMS created. | Assessments will be performed on baseline and 1 day after DOMS created.
  vertical jump test will be used for explosive power assessment
change between baseline of vertical jump test and 2 days after DOMS created. | Assessments will be performed on baseline and 2 days after DOMS created.
  vertical jump test will be used for explosive power assessment
change between baseline of vertical jump test and 3 days after DOMS created. | Assessments will be performed on baseline and 3 days after DOMS created.
  vertical jump test will be used for explosive power assessment
change between baseline of horizontal jump test and 1 day after DOMS created. | Assessments will be performed on baseline and 1 day after DOMS created.
  horizontal jump test will be used for explosive power assessment
change between baseline of horizontal jump test and 2 days after DOMS created. | Assessments will be performed on baseline and 2 days after DOMS created.
  horizontal jump test will be used for explosive power assessment
change between baseline of horizontal jump test and 3 days after DOMS created. | Assessments will be performed on baseline and 3 days after DOMS created.
  horizontal jump test will be used for explosive power assessment
change between baseline of thigh circumference measurement and immediately after DOMS created. | Assessments will be performed on baseline and immediately after DOMS created.
  Thigh circumference measurement will be used for thigh circumference assessment
change between baseline of thigh circumference measurement and 1 day after DOMS created. | Assessments will be performed on baseline and 1 day after DOMS created.
  Thigh circumference measurement will be used for thigh circumference assessment
change between baseline of thigh circumference measurement and 2 days after DOMS created. | Assessments will be performed on baseline and 2 days after DOMS created.
  Thigh circumference measurement will be used for thigh circumference assessment
change between baseline of thigh circumference measurement and 3 days after DOMS created. | Assessments will be performed on baseline and 3 days after DOMS created.
  Thigh circumference measurement will be used for thigh circumference assessment
change between baseline of Y balance test and 1 day after DOMS created. | Assessments will be performed on baseline and 1 day after DOMS created.
  Y balance test will be used for dynamic balance assessment
change between baseline of Y balance test and 2 days after DOMS created. | Assessments will be performed on baseline and 2 days after DOMS created.
  Y balance test will be used for dynamic balance assessment
change between baseline of Y balance test and 3 days after DOMS created. | Assessments will be performed on baseline and 3 days after DOMS created.
  Y balance test will be used for dynamic balance assessment

CONTACTS AND LOCATIONS:
Overall Officials: Erdoğan Çetintaş, PT, Principal Investigator — Eastern Mediterranean University; Berkiye Kırmızıgil, DPT, Study Director — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Mersin 10, Turkey, Cyprus

REFERENCES:
- [Background] Cheung K, Hume P, Maxwell L. Delayed onset muscle soreness : treatment strategies and performance factors. Sports Med. 2003;33(2):145-64. doi: 10.2165/00007256-200333020-00005. PMID 12617692
- [Background] Close GL, Ashton T, McArdle A, Maclaren DP. The emerging role of free radicals in delayed onset muscle soreness and contraction-induced muscle injury. Comp Biochem Physiol A Mol Integr Physiol. 2005 Nov;142(3):257-66. doi: 10.1016/j.cbpa.2005.08.005. Epub 2005 Sep 8. PMID 16153865
- [Background] Bleakley C, McDonough S, Gardner E, Baxter GD, Hopkins JT, Davison GW. Cold-water immersion (cryotherapy) for preventing and treating muscle soreness after exercise. Cochrane Database Syst Rev. 2012 Feb 15;2012(2):CD008262. doi: 10.1002/14651858.CD008262.pub2. PMID 22336838
- [Background] Bieuzen F, Bleakley CM, Costello JT. Contrast water therapy and exercise induced muscle damage: a systematic review and meta-analysis. PLoS One. 2013 Apr 23;8(4):e62356. doi: 10.1371/journal.pone.0062356. Print 2013. PMID 23626806
- [Background] Costello JT, Bieuzen F, Bleakley CM. Where are all the female participants in Sports and Exercise Medicine research? Eur J Sport Sci. 2014;14(8):847-51. doi: 10.1080/17461391.2014.911354. Epub 2014 Apr 25. PMID 24766579
- [Background] Jonhagen S, Ackermann P, Eriksson T, Saartok T, Renstrom PA. Sports massage after eccentric exercise. Am J Sports Med. 2004 Sep;32(6):1499-503. doi: 10.1177/0363546503262196. Epub 2004 Jul 20. PMID 15310577
- [Background] Johansson PH, Lindstrom L, Sundelin G, Lindstrom B. The effects of preexercise stretching on muscular soreness, tenderness and force loss following heavy eccentric exercise. Scand J Med Sci Sports. 1999 Aug;9(4):219-25. doi: 10.1111/j.1600-0838.1999.tb00237.x. PMID 10407930
- [Background] Donnelly AE, Maughan RJ, Whiting PH. Effects of ibuprofen on exercise-induced muscle soreness and indices of muscle damage. Br J Sports Med. 1990 Sep;24(3):191-5. doi: 10.1136/bjsm.24.3.191. PMID 2078806
- [Background] Baker RT, Hansberger BL, Warren L, Nasypany A. A NOVEL APPROACH FOR THE REVERSAL OF CHRONIC APPARENT HAMSTRING TIGHTNESS: A CASE REPORT. Int J Sports Phys Ther. 2015 Oct;10(5):723-33. PMID 26491622
- [Background] MacDonald N, Baker R, Cheatham SW. THE EFFECTS OF INSTRUMENT ASSISTED SOFT TISSUE MOBILIZATION ON LOWER EXTREMITY MUSCLE PERFORMANCE: A RANDOMIZED CONTROLLED TRIAL. Int J Sports Phys Ther. 2016 Dec;11(7):1040-1047. PMID 27999718
- [Background] Hammer WI. The effect of mechanical load on degenerated soft tissue. J Bodyw Mov Ther. 2008 Jul;12(3):246-56. doi: 10.1016/j.jbmt.2008.03.007. Epub 2008 Jun 3. PMID 19083680
- [Background] Lee JH, Lee DK, Oh JS. The effect of Graston technique on the pain and range of motion in patients with chronic low back pain. J Phys Ther Sci. 2016 Jun;28(6):1852-5. doi: 10.1589/jpts.28.1852. Epub 2016 Jun 28. PMID 27390432
- [Background] Markovic G. Acute effects of instrument assisted soft tissue mobilization vs. foam rolling on knee and hip range of motion in soccer players. J Bodyw Mov Ther. 2015 Oct;19(4):690-6. doi: 10.1016/j.jbmt.2015.04.010. Epub 2015 May 5. PMID 26592226
- [Background] Laudner K, Compton BD, McLoda TA, Walters CM. Acute effects of instrument assisted soft tissue mobilization for improving posterior shoulder range of motion in collegiate baseball players. Int J Sports Phys Ther. 2014 Feb;9(1):1-7. PMID 24567849
- [Background] Portillo-Soto A, Eberman LE, Demchak TJ, Peebles C. Comparison of blood flow changes with soft tissue mobilization and massage therapy. J Altern Complement Med. 2014 Dec;20(12):932-6. doi: 10.1089/acm.2014.0160. PMID 25420037
- [Background] Stroiney DA, Mokris RL, Hanna GR, Ranney JD. Examination of Self-Myofascial Release vs. Instrument-Assisted Soft-Tissue Mobilization Techniques on Vertical and Horizontal Power in Recreational Athletes. J Strength Cond Res. 2020 Jan;34(1):79-88. doi: 10.1519/JSC.0000000000002628. PMID 29742744
- [Background] Beardsley C, Skarabot J. Effects of self-myofascial release: A systematic review. J Bodyw Mov Ther. 2015 Oct;19(4):747-58. doi: 10.1016/j.jbmt.2015.08.007. Epub 2015 Aug 28. PMID 26592233
- [Background] Mikesky AE, Bahamonde RE, Stanton K, Alvey T, Fitton T. Acute effects of The Stick on strength, power, and flexibility. J Strength Cond Res. 2002 Aug;16(3):446-50. PMID 12173961
- [Background] MacDonald GZ, Penney MD, Mullaley ME, Cuconato AL, Drake CD, Behm DG, Button DC. An acute bout of self-myofascial release increases range of motion without a subsequent decrease in muscle activation or force. J Strength Cond Res. 2013 Mar;27(3):812-21. doi: 10.1519/JSC.0b013e31825c2bc1. PMID 22580977
- [Background] Sullivan KM, Silvey DB, Button DC, Behm DG. Roller-massager application to the hamstrings increases sit-and-reach range of motion within five to ten seconds without performance impairments. Int J Sports Phys Ther. 2013 Jun;8(3):228-36. PMID 23772339
- [Background] Bradbury-Squires DJ, Noftall JC, Sullivan KM, Behm DG, Power KE, Button DC. Roller-massager application to the quadriceps and knee-joint range of motion and neuromuscular efficiency during a lunge. J Athl Train. 2015 Feb;50(2):133-40. doi: 10.4085/1062-6050-49.5.03. Epub 2014 Nov 21. PMID 25415414
- [Background] Gajdosik RL, Bohannon RW. Clinical measurement of range of motion. Review of goniometry emphasizing reliability and validity. Phys Ther. 1987 Dec;67(12):1867-72. doi: 10.1093/ptj/67.12.1867. PMID 3685114
- [Background] Paschalis V, Nikolaidis MG, Theodorou AA, Giakas G, Jamurtas AZ, Koutedakis Y. Eccentric exercise affects the upper limbs more than the lower limbs in position sense and reaction angle. J Sports Sci. 2010 Jan;28(1):33-43. doi: 10.1080/02640410903334764. PMID 20013463